CLINICAL TRIAL: NCT01895062
Title: Effectiveness and Safety of Continuous Negative External Pressure (cNEP) in Preventing Sedation-Related Respiratory Impairment in Adults Undergoing Colonoscopy
Brief Title: Effectiveness of Continuous Negative External Pressure in Preventing Upper Airway Impairment During Routine Colonoscopy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: 5i Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5iS-009
Record Dates: First submitted 2013-03-29; First posted 2013-07-10 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Airway Obstruction; Apnea; Hypopnea
Keywords: colonoscopy; oxygen desaturation
MeSH Terms: conditions — Airway Obstruction; Apnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active cNEP @ -45cmw (Experimental): cNEP @ -45 cmw is applied to the anterior surface of the neck with a soft collar attached to a vacuum source.
  Interventions: Device: Airway Management System (AMS)
- no intervention (No Intervention): Routine care is administered without the application of cNEP.

INTERVENTIONS:
Device: Airway Management System (AMS) — The AMS consists of a silicone collar applied under the mandible to the anterior surface of the neck.
  The collar is attached to a vacuum source which delivers continuous negative external pressure to the upper airway.
  Arms: active cNEP @ -45cmw

SUMMARY:
The primary goal of this study is to determine the effectiveness and safety of delivering continuous negative external pressure (cNEP) to the upper airway as a means of preventing episodes of respiratory impairment (RI) such as hypoxemia, apnea and hypoventilation associated with the use of intravenous sedation in elective colonoscopy in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects undergoing elective colonoscopy at the Study Site who have fewer than three or more than three positive responses on the STOP BANG questionnaire

Exclusion Criteria:

* Presence of severe cardiopulmonary or neurologic disease as determined by the investigator
* History of vascular fragility associated with cutaneous pressure
* History of hypersensitivity to silicone
* Inability to properly fit cNEP collar to the subject
* The presence of excessive facial hair in the region where the cNEP collar is positioned
* Known carotid vascular disease, previous major neck surgery or radiation therapy to the cervical region
* Presence of anatomical abnormalities in the neck or pharyngeal region (such as enlarged tonsils)
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Coyle, M.D., Principal Investigator — Scripps Healthcare
Locations (1):
- Scripps Green Clinic, La Jolla, California, United States

REFERENCES:
- [Derived] Kais SS, Klein KB, Rose RM, Endemann S, Coyle WJ. Continuous negative external pressure (cNEP) reduces respiratory impairment during screening colonoscopy: a pilot study. Endoscopy. 2016 Jun;48(6):584-7. doi: 10.1055/s-0042-102533. Epub 2016 Apr 25. PMID 27110692

RESULTS

PARTICIPANT FLOW:
Groups:
- Active cNEP @ -45cmw: cNEP @ -45 cmw is applied to the anterior surface of the neck with a soft collar attached to a vacuum source.
  Airway Management System (AMS): The AMS consists of a silicone collar applied under the mandible to the anterior surface of the neck.
  The collar is attached to a vacuum source which delivers continuous negative external pressure to the upper airway.
Period: Overall Study
Arm/Group | Active cNEP @ -45cmw | no Intervention
Started | 30 | 24
Completed | 30 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants in the cNEP group was estimated from the number required to show a 50% decrease in the primary endpoint compared to the no intervention group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active cNEP @ -45cmw | no Intervention | Total
Number analyzed (Participants) | 30 | 24 | 54
Age, Continuous [Mean (Full Range); unit: years] | 60 [33 to 78] | 60 [34 to 77] | 60 [33 to 78]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 18 | 40
  >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 27
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 30 | 24 | 54
History of sleep apnea [Number; unit: participants] — history of sleep apnea as reported by the study participant
  participants | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: RI Events in the cNEP Group Compared to the no cNEP Group, Where RI is Defined as Either: i Oxygen Saturation < 90% or ii. Apneas/Hypopneas of > 15 Sec Duration i. Oxygen Saturation <90% ii. Presence of Apneas or Hypopneas
Description: Mean RI events in the no cNEP group was 3.5 compared to 1.92 in the cNEP group (p=0.022)
Time Frame: 1 hour
Population: Not all subjects were evaluable due to malfunction of the respiratory monitoring equipment in several.
Measure: Mean (95% Confidence Interval); unit: RI events
Arm/Group | Active cNEP @ -45cmw | no Intervention
Number analyzed (Participants) | 29 | 24
RI events | 1.92 [1.1 to 2.75] | 3.5 [2.37 to 4.64]
Statistical Analysis 1: Comparison: Active cNEP @ -45cmw vs no Intervention; Test type: Superiority or Other; p < 0.022, t-test, 2 sided

2. Secondary Outcome: The Safety of cNEP as Determined by Adverse Events Reported by the Investigators.
Time Frame: 1 hour
Reporting Status: Not Posted

3. Secondary Outcome: The Incidence of Subjects With One or More RI in the cNEP Group Compared to the no cNEP Group.
Time Frame: 1 hour
Reporting Status: Not Posted

4. Secondary Outcome: The Frequency of Interventions to Alleviate RI in the cNEP Group Compared to the no cNEP Group.
Description: interventions such as reduction of sedative medication or jaw thrust.
Time Frame: 1 hour
Measure: Number; unit: interventions to restore airway
Arm/Group | Active cNEP @ -45cmw | no Intervention
Number analyzed (Participants) | 29 | 24
interventions to restore airway | 1 | 0

ADVERSE EVENTS:
Arm/Group | Active cNEP @ -45cmw | no Intervention
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/24
Other Adverse Events (participants affected / at risk) | 0/30 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No